CLINICAL TRIAL: NCT00976118
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group Study to Evaluate the Efficacy of Oral AB1010 in Adults Patients With Mild to Moderate Alzheimer-type Disease.
Brief Title: Activity of Masitinib (AB1010) in Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB04024
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Alzheimer's Disease
Keywords: Dementia of Alzheimer's type; mild to moderate Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- oral masitinib (AB1010) (Experimental): masitinib (AB1010) 3 or 6 mg/kg/day
  Interventions: Drug: masitinib (AB1010)

INTERVENTIONS:
Drug: masitinib (AB1010) — oral masitinib 3 or 6 mg/kg/day
  Other Names: AB1010
  Arms: oral masitinib (AB1010)
Drug: placebo — matching placebo to masitinib
  Arms: placebo

SUMMARY:
This phase 2 study was designed to evaluate the activity of oral masitinib (AB1010) administered at 2 dose levels during 24 weeks to patients with mild to moderate confirmed Alzheimer's type disease.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients from both sex
2. Age ≥ 50 years at screening
3. Menopause ≥ 2 years for women
4. Dementia of Alzheimer's type, according to DSM IV criteria
5. Probable Alzheimer' disease according to NINCDS-ADRDA criteria
6. MMSE ≥ 12 and ≤ 26 at baseline
7. CDR of 1 or 2 at baseline
8. Treated for a minimum of 6 months with a stable dose of cholinesterase inhibitors (donepezil, rivastigmine or galantamine) at baseline, and/or a stable dose of memantine for a minimum of 3 months at baseline, with no changes foreseen in therapy throughout the study
9. Presence of a reliable caregiver
10. Patient, identified caregiver and, if applicable, patient surrogate are able and willing to comply with study visits and procedures per protocol, understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed
11. Affiliated to the French Social Security regimen

Exclusion Criteria:

1. Any cause of dementia not due to Alzheimer's disease :

   * other central nervous conditions causing progressive deficits in memory and cognition, e.g. cerebrovascular disease, Parkinson's disease, Huntington's disease, brain tumor…
   * systemic conditions known to cause dementia, e.g., hypothyroidism, untreated vitamin B12 or folic acid deficiency, niacin deficiency, neurosyphilis, HIV infection…
   * substance-induced conditions
2. Alzheimer disease with delusions or delirium
3. Treatment with any registered or putative cognitive enhancer or disease modifier other than donepezil, galantamine, rivastigmine or memantine
4. Uncontrolled depression at screening
5. Evidence of psychosis and/or use of antipsychotic drugs at screening, or history of significant psychotic disorder or hospitalization for psychiatric disorders
6. Active current bacterial, viral (including hepatitis B and C, HIV, EBV, CMV, herpes zoster, herpes simplex), fungal, mycobacterium, protozoan, or other infection.
7. History of infection requiring hospitalization or treatment with antibiotics within 2 weeks of screening
8. Inadequate organ function, defined as follows : total bilirubin ≥ 1.5 x ULN, SGOT and SGPT ≥ 2.5 x UNL, creatinine clearance calculated by Crocroft method < 35 ml/mn, ANC ≤ 2500, platelets ≤ 100 000 at baseline
9. Treatment with any investigational agent within 4 weeks of screening,
10. Men and their partner refusing to use 2 methods of medically acceptable forms of contraception during the study.
11. History of poor compliance or history of drug/alcohol abuse, or excessive alcohol beverage consumption that would interfere with the ability to comply with the study protocol, or current or past psychiatric disease that might interfere with the ability to comply with the study protocol or give informed consent
12. Any condition that, in the investigator's opinion, could be detrimental to subjects participating in this study as life expectancy < 1 year, or any clinically important deviations from normal clinical laboratory values or concurrent medical events.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
change from baseline in ADAS-Cog | week 24

SECONDARY OUTCOMES:
change from baseline in CIBIC-plus | week 24
change from baseline in CDR | week 24
change from baseline in MMSE | week 24

REFERENCES:
- [Result] Piette F, Belmin J, Vincent H, Schmidt N, Pariel S, Verny M, Marquis C, Mely J, Hugonot-Diener L, Kinet JP, Dubreuil P, Moussy A, Hermine O. Masitinib as an adjunct therapy for mild-to-moderate Alzheimer's disease: a randomised, placebo-controlled phase 2 trial. Alzheimers Res Ther. 2011 Apr 19;3(2):16. doi: 10.1186/alzrt75. PMID 21504563
- See also: Publication of results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3226277/